CLINICAL TRIAL: NCT05330923
Title: Screening and Follow-up in Patients With HIV Infection Combined With Metabolic Associated Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Wuxi Hisky Medical Technology Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH record HS-3401D
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Fibrosis; HIV/AIDS
Keywords: integrase inhibitors; non-nucleoside reverse transcriptase inhibitors; transient elastography; iLivTouch
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identifying patients at risk of NAFLD(Nonalcoholic fatty liver disease), especially severe disease with NASH(nonalcoholic steatohepatitis) and fibrosis, is critical. Prevalence of NAFLD in PLWH(People Living With HIV) evaluated by different imaging techniques including US (ultrasonography), elastography, CT(computed tomography ), and magnetic resonance varies from 13% to 58.6% in all published studies. In previous studies, the effect of ART(Anti-Retroviral Therapy) on NAFLD was limited. A cross-sectional analysis found that INSTI（Integrase strand transfer inhibitor） was associated with a higher prevalence of steatosis in AIDS (acquired immunodeficiency syndrome) patients. However, it is not clear whether there is a difference in the degree of nonalcoholic steatosis between AIDS patients receiving NNRTI(non-nucleoside reverse transcriptase inhibitors).

Therefore, the investigators plan to conduct a prospective study to assess whether there is any difference in the degree of nonalcoholic steatosis and fibrosis between Chinese HIV(human immunodeficiency virus)/AIDS patients after initial treatment with NNRTI or INSTI, or switching from NNRTI to INSTI.

DETAILED DESCRIPTION:
Chronic liver disease is now a leading cause of non-AIDS-related death, representing 13% of all deaths in this patient population. While coinfection with viral hepatitis is the primary cause of liver disease, hepatic steatosis is emerging as a major contributor. NAFLD is defined by liver steatosis, the accumulation of triglycerides in the hepatocytes, in the absence of a secondary cause such as excessive alcohol consumption. The condition encompasses a spectrum of diseases from nonalcoholic fatty liver to NASH, fibrosis and cirrhosis. Recent studies report a wide range of prevalence of NAFLD between 15% and 60% among HIV patients. In non-HIV patients NAFLD is principally the hepatic manifestation of the metabolic syndrome, occurring in the context of insulin resistance, central obesity and dyslipidaemia, with disease progression involving a number of complex interacting factors such as genetic susceptibility, oxidative stress and dysbiosis. There is a growing body evidence for weight gain following initiating integrase inhibitor therapy, particularly with dolutegravir and bictegravir. However, the consequences of weight gain have not been evaluated.

Identifying patients at risk of NAFLD, especially severe disease with NASH and fibrosis, is critical. Prevalence of NAFLD in PLWH evaluated by different imaging techniques varies from 13% to 58.6% in all published studies. In previous studies, the effect of ARTon NAFLD was limited. A cross-sectional analysis found that INSTI was associated with a higher prevalence of steatosis in AIDS patients. However, it is not clear whether there is a difference in the degree of nonalcoholic steatosis between AIDS patients receiving NNRTI.

Transient elastography is a non-invasive technique to measure UAP(ultrasound attenuation parameter)and liver stiffness simultaneously. The former reflects the degree of hepatic steatosis. The typical features of fatty liver on abdominal ultrasonography include bright liver echotexture, deep attenuation of ultrasound signal and vascular blunting. The latter two features are because of the faster attenuation of ultrasound wave amplitude in a steatotic liver. UAP takes advantage of this physical property and estimates the ultrasound attenuation at the central frequency of transient elastography, while assuming a homogeneous fat distribution and an adequate penetration.

Therefore, the investigators plan to conduct a prospective study to assess whether there is any difference in the degree of nonalcoholic steatosis and fibrosis between Chinese HIV/AIDS patients after initial treatment with NNRTI or INSTI, or switching from NNRTI to INSTI.

ELIGIBILITY:
Inclusion Criteria:

* Newly treated or treated AIDS patients;
* Regular follow-up visits to the hospital, medication compliance is good;
* Patients or their family members were willing to participate in the study by understanding the study plan and providing written informed consent.

Exclusion Criteria:

* Unable to complete the position requirements of ultrasonic examination (lying flat) due to mobility difficulties;
* Patients have poor compliance and cannot follow up regularly or take medicine on time;
* Patients or family members cannot understand the conditions and objectives of the study;
* Other conditions considered unsuitable for inclusion by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly treated or treated AIDS patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
The degree of hepatic steatosis and fibrosis | 12 months
  The ultrasound attenuation parameter(UAP) and liver stiffness in HIV/AIDS patients treated with either of INSTI and NNRTI for at least 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: WEI Lyu, Principal Investigator — Department of Infectious Diseases, PekingUMCH
Locations (1):
- Chinese Academy of Medical Sciences Peking Union Medical College Hospital, Beijing, Beijing Municipality, China